CLINICAL TRIAL: NCT00594854
Title: 6-Month, Randomized, Double-blind, Parallel-group, Controlled, Multi-center Study of Gastric Ulcer Incidence With PN400 (Esomeprazole/Naproxen) Versus Diclofenac/Misoprostol in Subjects at High Risk for Developing NSAID-Associated Ulcers
Brief Title: Evaluating PN 400 (VIMOVO) in Reducing Gastric Ulcers in High Risk Subjects Compared to Arthrotec
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: POZEN agreed with FDA to stop study due to low and inadequate enrollment
Sponsor: POZEN (Industry)
Responsible Party: Everardus Orlemans, PhD, VP, Clinical Research, POZEN Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN400-303
Record Dates: First submitted 2007-12-19; First posted 2008-01-16 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-08

CONDITIONS: Gastric Ulcer
Keywords: NSAID; Gastric Ulcer; High risk; Arthrotec; Vimovo
MeSH Terms: conditions — Stomach Ulcer | interventions — Arthotec; Arthrotec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PN400 (Experimental): PN 400 (esomeprazole/naproxen) dosed twice daily
  Interventions: Drug: PN400 (VIMOVO)
- Diclofenac/Misoprostol (Active Comparator): diclofenac 75mg/misoprostol 200 mcg dosed twice daily
  Interventions: Drug: Diclofenac/Misoprostol

INTERVENTIONS:
Drug: PN400 (VIMOVO) — PN400 tablet (500 mg delayed-release naproxen/20 mg immediate-release esomeprazole) given by mouth twice daily (bid).
  Other Names: Vimovo
  Arms: PN400
Drug: Diclofenac/Misoprostol — Over-encapsulated ARTHROTEC® 75 (75 mg diclofenac sodium/200 mcg misoprostol) capsules given by mouth bid.
  Other Names: Arthrotec
  Arms: Diclofenac/Misoprostol

SUMMARY:
This randomized, double-blind, parallel-group, controlled, multi-center clinical trial of 6 months duration is designed to assess the efficacy, tolerability and safety of PN400 versus diclofenac/misoprostol in subjects at high risk for developing NSAID-associated gastric ulcers. Approximately 100 sites will participate to enroll a total of 200 subjects (100 per arm).

At least 20% of the subjects enrolled will be age 65 years and older.

DETAILED DESCRIPTION:
To determine the incidence of gastric ulcers following administration of PN 400 in a high risk population over six months. Diclofenac/misoprostol will be used as a positive control.

Secondary:

* To determine the incidence of duodenal ulcers during treatment with PN 400 and diclofenac/misoprostol in a high risk population
* To evaluate the degree of upper gastrointestinal injury as measured by Lanza scores (1991) during treatment with PN400 and diclofenac/misoprostol in a high risk population
* To compare gastrointestinal symptoms in subjects treated with PN 400 versus diclofenac/misoprostol as measured by scores on the Gastrointestinal Symptoms Rating Scale (GSRS) instrument
* To evaluate the safety and tolerability of PN400 and diclofenac/misoprostol in a high risk population

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female subjects, 18 years and older with a history of osteoarthritis, rheumatoid arthritis, ankylosing spondylitis or other medical condition expected to require daily NSAID therapy for at least 6 months, with a documented history of an ulcer related serious upper gastrointestinal event such as bleeding, perforation or obstruction
2. Female subjects are eligible for participation in the study if they are of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant);
   * Childbearing potential, have a negative pregnancy test at screening, and at least one of the following applies or is agreed to by the subject:

     * Female sterilization or sterilization of male partner; or,
     * Hormonal contraception by oral route, implant, injectable, vaginal ring; or,
     * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year;
     * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide); or
     * Any other method with published data showing that the lowest expected failure rate is less than 1% per year
3. Each subject must be able to understand and comply with study procedures required of a subject and is able and willing to provide written informed consent prior to any study procedures being performed

Exclusion Criteria:

1. History of hypersensitivity to esomeprazole or to another proton-pump inhibitor
2. History of allergic reaction or intolerance to any NSAID (including aspirin) and/or a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps
3. Positive test result for H. pylori at screening
4. Participation in any study of an investigational treatment in the 4 weeks before screening
5. Presence of uncontrolled acute or chronic medical illness, e.g. gastrointestinal disorder, hypertension, diabetes, thyroid disorder, depression and/or infection that would endanger a subject if they were to participate in the study
6. Gastrointestinal disorder or surgery leading to impaired drug absorption
7. Evidence of uncontrolled, or unstable cardio- or cerebrovascular disorder, which in the investigator's opinion would endanger a subject if they were to participate in the study
8. Schizophrenia or bipolar disorder
9. Use of any excluded concomitant medication (see Section 9.2)
10. A recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence, including overuse/abuse of narcotics for management of pain
11. Serious blood coagulation disorder, including use of systemic anticoagulants
12. Screening endoscopy showing >10 erosions or any gastric or duodenal ulcer at least 3 mm in diameter with depth
13. Screening laboratory ALT or AST value > 2 times the upper limit of normal
14. Estimated creatinine clearance < 50 ml/min
15. Other than noted specifically, any screening laboratory value that is clinically significant in the investigator's opinion and would endanger a subject if they were to participate in the study
16. History of malignancy, treated or untreated, within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everardus Orlemans, PhD, Study Chair — POZEN
Locations (1):
- POZEN, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-center US study, 16 sites recruited subjects between November 2007 and June 2008. On May 2, 2008 POZEN reached agreement with the FDA to terminate the study based on difficulty in recruiting subjects.
Pre-assignment Details: Screening for eligibility and wash-out of restricted medications.
Groups:
- PN400 (VIMOVO): PN 400 (esomeprazole/naproxen) dosed twice daily (bid)
- Arthrotec: diclofenac/misoprostol dosed twice daily (bid)
Period: Overall Study
Arm/Group | PN400 (VIMOVO) | Arthrotec
Started | 9 | 11
Completed | 2 (POZEN reached an agreement with the FDA to terminate the study due to low and inadequate enrollment.) | 1 (POZEN reached an agreement with the FDA to terminate the study due to low and inadequate enrollment.)
Not Completed | 7 | 10
Not completed — Study terminated | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PN400 (VIMOVO) | Arthrotec | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.5) | 54.4 (17.2) | 58.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Duodenal Ulcers Confirmed by Endoscopy
Description: Number of participants with duodenal ulcers confirmed by endoscopy following administration of PN 400 VIMOVO)or Arthrotec in a high risk population
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | PN400 (VIMOVO) | Arthrotec
Number analyzed (Participants) | 9 | 11
participants | 0 [0 to 33.6] | 1 [0.2 to 41.3]

2. Primary Outcome: Number of Participants With Gastric Ulcer Confirmed by Endoscopy
Description: Number of participants with gastric ulcers confirmed by endoscopy following administration of PN 400 (VIMOVO) or Arthrotec in a high risk population over six months.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | PN400 (VIMOVO) | Arthrotec
Number analyzed (Participants) | 9 | 11
Participants | 2 | 1

3. Secondary Outcome: Number of Participants With Upper Gastro-intestinal Injury Grade 4 as Measured by Lanza (1991) Score
Description: The degree of upper gastrointestinal (UGI) injury as measured by Lanza scores (1991) during treatment with PN 400 and ARTHROTEC® in a high-risk population. The Lanza (1991) score is based on endoscopic obeservations and rating these, with no damage, petecchiae, erosions and ulcers. On the 1991 scale, a Lanza score of 0 represents normal mucosa (no damage), while a score of 4 indicates 6-10 erosions, and a score of 7 indicates an ulcer.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | PN400 (VIMOVO) | Arthrotec
Number analyzed (Participants) | 9 | 11
participants | 2 [0 to 0] | 2 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data collection were planned at 1, 3 and 6 months. In May 2008 POZEN reached an agreement with the FDA to terminate the study due to low and inadequate enrollment. No 6 month adverse events data were collected.
Arm/Group | PN400 (VIMOVO) | Arthrotec
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 7/9 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN400 (VIMOVO) (N=9) | Arthrotec (N=11)
Gastritis Erosive (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less